CLINICAL TRIAL: NCT03670563
Title: Training Intrinsic Foot Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Katherine Newsham PhD, ATC, Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 29267
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Muscular Weakness
Keywords: Therapeutic exercise
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two intervention arms and one control arm
Who Masked: Outcomes Assessor
Masking Description: Team members collecting outcomes data will not know participant allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise 1 (Experimental): Short foot exercise protocol instructed utilizing verbal instruction, passive modeling, active-assisted modeling, and active modeling.
  Interventions: Other: Short foot exercise protocol
- Exercise 2 (Active Comparator): Short foot exercises plus NMES. Short foot exercise protocol instructed utilizing verbal instruction, passive modeling assisted by neuromuscular electric stimulation (NMES), active-assisted modeling assisted by neuromuscular electric stimulation, and active modeling.
  Interventions: Other: Short foot exercise plus NMES
- Control (No Intervention): No exercise intervention; continue normal physical activity, but do not start any new exercise programs

INTERVENTIONS:
Other: Short foot exercise protocol — Exercises that target intrinsic foot muscles
  Arms: Exercise 1
Other: Short foot exercise plus NMES — Exercises that target intrinsic foot muscles supplemented by NMES for muscle re-education
  Arms: Exercise 2

SUMMARY:
The foot intrinsic muscles are increasingly targeted in foot and ankle rehabilitation. The exercises are often difficult to learn initially. The purpose of the proposed study is to examine the effect training the intrinsic foot muscles on performance in selected physical and functional measures such as balance, plantar pressure during gait, vertical jump, and foot posture. In addition,the investigators will compare one group training with traditional exercise instruction methods and one group using an adjunctive modality (neuromuscular electric stimulation) during the introductory phases of exercise instruction. The investigators are interested in how this modality might affect physical and functional outcome measures and if it affects participants' frustration with learning a new exercise.

DETAILED DESCRIPTION:
Arm 1: The purpose of this arm of the study is to determine if a 4-week trial of foot muscle exercises, instructed with passive, active-assisted, and active techniques, affect functional measures such as balance, plantar pressure during gait, and vertical jump. A frustration index will be employed to assess participant frustration with learning a new exercise. 15 will be enrolled in this arm of the study.

Arm 2: The purpose of this arm of the study is to determine if a 4-week trial of foot muscle exercises, instructed with neuromuscular electric stimulation (NMES) and active techniques, affect functional measures such as balance, plantar pressure during gait, and vertical jump. A frustration index will be employed to assess participant frustration with learning a new exercise.15 will be enrolled in this arm of the study.

Arm 3: This group will not engage in any training, but will serve as a comparator for the two intervention arms.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-30; Participate in physical activity 3 times/week; No neurologic injury/condition; No prior experience with study exercises; No injury to lower extremity in past 2 months; Inability to selectively extend the great toe while the lesser toes remain quiet (indicating INTRINSIC FOOT MUSCLES dysfunction)

Exclusion Criteria:

* Sedentary; Known neurologic injury or condition; Current LE injury that may affect neuromuscular function; Tarsal coalition; Absolute contradiction to manual therapy or neuromuscular electrical stimulation (NMES); Previous intrinsic foot muscle training protocol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Reaching Distance | Arm 1 and Arm 2: Baseline, 2 weeks, 4 weeks, 8 weeks. Arm 3: Baseline 4 weeks, 8 weeks
  The change demonstrated in clinical test of single limb reach/balance in the anterior, posterolateral, and posteriomedial directions in cm
Center of pressure during walking gait | Arm 1 and Arm 2: Baseline, 2 wk, 4 wk, 8 wk. Arm 3: Baseline 4 wk, 8 wk
  Changes in center of pressure during walking gait

SECONDARY OUTCOMES:
Changes in foot posture over loading conditions | Arm 1 and Arm 2: Baseline, 2 weeks, 4 weeks, 8 weeks. Arm 3: Baseline 4 weeks, 8 weeks
  Change in navicular height from 10% weight bearing to 90% weight bearing in mm
Arch Height Index | Arm 1 and Arm 2: Baseline, 2 weeks, 4 weeks, 8 weeks. Arm 3: Baseline 4 weeks, 8 weeks
  Change in arch height from 10% weight bearing to 90% weight bearing relative to truncated foot length (in %)
Maximal vertical jump height | Arm 1 and Arm 2: Baseline, 2 weeks, 4 weeks, 8 weeks. Arm 3: Baseline 4 weeks, 8 weeks
  Maximal height jump off of two feet will be measured in centimeters
Changes in landing forces | Arm 1 and Arm 2: Baseline, 2 weeks, 4 weeks, 8 weeks. Arm 3: Baseline 4 weeks, 8 weeks
  Change in vertical ground reaction force during landing after vertical jump
Perceived effort in learning novel exercise measured by NASA-Task Load Index (NASA-TLX) | Arm 1 and Arm 2: Supervised training sessions 1, 2, 3, 4, 5, and 6
  Participant reported workload estimates of Mental, Physical, and Temporal Demands, Frustration, Effort, and Performance. RAW TLX will be utilized, with each component considered individually; the subscales will not be combined. Subscales are rated 0-21; higher scores indicate greater load or difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Newsham, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No